CLINICAL TRIAL: NCT04090866
Title: Cardiac Metabolic Remodeling After Pulmonary Vasodilator Therapy in Pulmonary Arterial Hypertension: A Pilot Study
Status: Terminated | Type: Observational
Why Stopped: PI and sponsor will re-open study at new institution, will not transfer data due to COVID-19 situation
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: 2019-0286; A534285 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*P (Other: UW Madison); Protocol Version 8/2/2019 (Other: UW Madison)
Record Dates: First submitted 2019-09-12; First posted 2019-09-16 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Arterial Hypertension; Right-Sided Heart Failure
Keywords: pulmonary arterial hypertension; right-sided heart failure; metabolism; PET/MRI
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PET/MRI — Positron Emission Tomograph/Magnetic Resonance Imaging - participants will undergo PET/MRI prior to initiation of pulmonary vasodilator therapy and again 4-6 months after initiation of therapy

SUMMARY:
Pulmonary arterial hypertension(PAH) is associated with the development of right heart failure. In the setting of heart failure, the heart shifts to increasing dependence on glucose metabolism. In this study, the investigators will perform cardiac positron emission tomography/magnetic resonance imaging (PET/MRI) scans to measure glucose metabolism in the heart before and after initiation of pulmonary vasodilator therapy for pulmonary arterial hypertension.

DETAILED DESCRIPTION:
Pulmonary arterial hypertension is associated with the development of right heart failure. In the setting of heart failure, the heart shifts to increasing dependence on glucose metabolism. In this study, the investigators will perform cardiac positron emission tomography/magnetic resonance imaging (PET/MRI) scans to measure glucose metabolism in the heart before and after initiation of pulmonary vasodilator therapy for pulmonary arterial hypertension. By utilizing a rest-exercise protocol and continuous PET imaging acquisition, we can capture real-time changes in glucose uptake in the heart in response to acute exercise. By coupling these measures of dynamic glucose utilization with MRI-based cardiac function, we will determine cardiac metabolic efficiency.

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization(WHO) group PAH secondary into idiopathic pulmonary arterial hypertension(IPAH) or connective tissue disease associated pulmonary arterial hypertension (CTDPAH)
* New York Heart Association (NYHA) classification I - III heart failure
* Vasodilator therapy naive
* Able to provide informed consent

Exclusion Criteria:

* Metabolic disorders such as uncontrolled diabetes (A1c > 8%) that may interfere with FDG uptake
* Baseline 6-minute walk distance (6MWD) < 400 feet or NYHA class IV heart failure
* Musculoskeletal abnormalities that would prevent exercise
* Contraindications to MRI

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IPAH or CTD-PAH
Sampling Method: Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-07-21 (Actual)

PRIMARY OUTCOMES:
Ability to augment glucose uptake ("substrate flexibility"), defined as change in rate of glucose uptake from rest to exercise | 6 months
  Substrate flexibility is defined as the change in myocardial to blood pool glucose uptake rate from rest to exercise.

SECONDARY OUTCOMES:
Change in substrate flexibility after initiation of pulmonary vasodilator therapy | 6 months
  Substrate flexibility is defined as the change in myocardial to blood pool glucose uptake rate from rest to exercise. Substrate flexibility before and after pulmonary vasodilator therapy will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Kara Goss, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin-Madison, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No